

# Visual Outcomes, Patient Satisfaction and Spectacle Independence Evaluation of the Acrysof® IQ Vivity® Intraocular Lens Targeted for Emmetropia or Nanovision.

| Sponsor: | Carolina Eyecare Physicians, LLC<br>1101 Clarity Rd., Suite 100<br>Mt. Pleasant, SC 29466<br>(843) 881 3937<br>Kerry D. Solomon, MD, Principal Investigate<br>Helga P. Sandoval, MD, MSCR, Director of F | |
|---|---|---|
| Study Product: | AcrySof® IQ Vivity (DAT015 and DATx15) in | traocular lenses |
| Protocol Number: | CEP-20-002<br>Initial version date: 22April2020 | |
| Investigator Agreement: | I have read the clinical study described herein, recognize its confidentiality and agree to conduct the described trial in compliance with Good Clinical Practices (GCP), the Declaration of Helsinki, this protocol and all applicable regulatory requirements. Additionally, I will comply with all procedures for obtaining informed consent, data recording and reporting, will permit monitoring, auditing, and inspection of my research center, and will retain all records until notified by the sponsor. | |
| Name of the Investigator:<br>Name of the Institution:<br>Address: | | |
| Principal Investigator: | <del></del> | |
| | Signature | Date |



# Visual Outcomes, Patient Satisfaction and Spectacle Independence Evaluation of the Acrysof® IQ Vivity® Intraocular Lens Targeted for Emmetropia or Nanovision.

Current visual outcomes expectations of cataract patients are similar to those of refractive surgery patients. Their desire is to be spectacle independent for far, intermediate and near vision activities. Some may have already enjoyed freedom from glasses and would like to continue after the cataracts are removed. Different options are available. These options include mono-vision and presbyopia correcting intraocular lenses (IOL).

Presbyopia correcting IOLs include accommodative, multifocals, extended depth of focus (EDOF) and trifocal IOLs.

Multifocal IOLs (MIOLs) were FDA approved in 1997 and have been classified based on their design as refractive or diffractive. Refractive MIOLs (i.e ReZoom) reportedly provided better intermediate vision while diffractive MIOLs (i.e ReSTOR) provided better near visual acuity. Mixing and matching these lenses was an option to overcome the limitations each one presented providing patients improved intermediate and near acuities. The ReSTOR was modified and the ReZoom IOL was discontinued.

The original ReSTOR has a +4.0 D add with good uncorrected distance and near visual acuities (UCDVA, UCNVA) with a reading distance of 33 cm but with limited intermediate acuity. Two additional ReSTOR models are currently available, a +3.0 D add to enhance the intermediate distance vision with a reading distance of 40 cm, and a +2.5 D add ideal for people who are interested in distance and intermediate vision (50 - 60 cm) activities. One potential disadvantage of the low add multifocal IOLs is the visual performance at near. Similarly, to mixing and matching, the use of a ReSTOR +3.0 in one eye and the +2.5 in the fellow eye, known as blended vision, is an option to improve patients' vision at the different distances reducing their dependence on glasses.

Another option to manage this potential shortcoming is to set the non-dominant eye for a small residual myopic error (-0.50 D) what is referred to as mini mono-vision or nanovision. A previous study evaluating the visual outcomes of the Symfony Toric IOL when both eyes were targeted for emmetropia and when the non-dominant eye was targeted for nano-vision (-0.50 D) in patients with astigmatism showed that the nanovision approach provided similar binocular acuity at distance and intermediate but better acuity at near with high patient satisfaction and less dependence on glasses.

In August 2019, the FDA approved the first trifocal in USA. The PanOptix trifocal IOL provides excellent vision at all 3 distances with about 92% of patients near VA at 40 cm was 20/25 or better while at 66 cm, 94% were 20/25 or better overcoming the "weakness" of previous presbyopia correcting IOLs.

3

However, patients' complaints of glare, halos and starburst are common with all this type of lenses. The severity of these visual symptoms varies according to the actual IOL design.

The recently approved Vivity Extended Vision IOL is not a multifocal IOL but due to its design, it provides better intermediate and near VA compared to a monofocal IOL. Reported visual disturbances are comparable to those reported by patients implanted with monofocal lenses which are less than those reported by patients implanted with multifocal or extended depth of focus lenses.

# 1. OBJECTIVE:

The purpose of this study is to evaluate the visual outcomes and defocus curve, visual disturbances, patient satisfaction and spectacle independence of the AcrySof® IQ Vivity® IOL when both eyes are targeted for emmetropia and when the non-dominant eye is targeted for nano-vision (-0.50D) in patients with or without astigmatism after routine cataract surgery.

# 2. STUDY ENDPOINTS:

# 1. Primary Endpoints:

a. Binocular uncorrected<sup>†</sup> near (40 cm) visual acuity

# 2. Secondary Endpoints:

- a. Binocular distance-corrected near (40 cm) visual acuity at 3 months
- b. Binocular uncorrected and distance-corrected intermediate (66 cm) visual acuity at 3 months
- c. Binocular uncorrected and best-corrected distance (4 m) visual acuity at 3 months
- d. Binocular defocus curve at 3 months
  - Will be performed with both eyes set for plano
  - Will be performed with dominant eye set for plano and non-dominant eye set for -0.50D
- e. To evaluate patient's vision satisfaction at 3 months (Intraocular Lens Satisfaction IOLSAT)
- f. To evaluate patient's spectacle independence 3 months (IOLSAT)
- g. To evaluate visual symptoms using a questionnaire 3 months (Questionnaire for Visual Disturbance (QUVID)

# 3. STUDY DESIGN:

Prospective, single center, non-randomized, bilateral eye study. In all subjects, the target refraction for the dominant eye will be plano (±0.25 D) and between -0.50 and -0.75 D (closest to -0.62) for the non-dominant eye. At the postoperative visit, subjects will be evaluated twice. One time with both eyes correct for plano (target emmetropia) and the second time the dominant eye will be corrected for plano and the non-dominant eye for -0.50 (target nanovision). Subjects will be randomized to

which target is evaluated first (i.e. First evaluation: Target emmetropia – Second evaluation: Target nanovision or First evaluation: Target nanovision – Second evaluation: Target emmetropia. There will be a 10-minute break between evaluations.

4

#### 4. INCLUSION/EXCLUSION CRITERIA

#### 4.1. Inclusion Criteria:

Subjects MUST fulfill the following conditions to qualify for enrollment into the trial

- 1. Subject is undergoing bilateral lens extraction with intraocular lens implantation.
- 2. Gender: Males and Females.
- 3. Age: 50 years and older.
- 4. Willing and able to provide written informed consent for participation in the study
- 5. Willing and able to comply with scheduled visits and other study procedures.
- 6. Scheduled to undergo standard cataract surgery with topical anesthesia in both eyes within 6 to 30 days between surgeries
- 7. Subjects who require an IOL power in the range of +15.0 D to +25.0 D only.
- 8. Subjects who require a toric IOL up to +3.00 D at the IOL plane (2.06 D corneal plane).
- 9. Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

#### 4.2. Exclusion Criteria:

Subjects with <u>ANY</u> of the following conditions on the eligibility exam may <u>NOT</u> be enrolled into the trial.

- 1. Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
- 2. Uncontrolled diabetes.
- 3. Use of any systemic or topical drug known to interfere with visual performance.
- 4. Contact lens use during the active treatment portion of the trial.
- 5. Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
- 6. Clinically significant corneal dystrophy
- 7. History of chronic intraocular inflammation.
- 8. History of retinal detachment.
- 9. Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
- 10. Previous intraocular surgery.
- 11. Previous corneal refractive surgery (i.e. LASIK, PRK, RK).
- 12. Previous keratoplasty

5

- 13. Severe dry eye
- 14. Pupil abnormalities
- 15. Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
- 16. Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
- 17. Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates the patient is unsuitable for the trial.

# 4.3. Exclusion Criteria at time of surgery:

If any of the following exclusion criteria are applicable to the study eye, the subject should not continue in the study.

- 1. Other ocular surgery procedures, i.e. iStent, anterior vitrectomy
- 2. Significant vitreous loss
- 3. Significant anterior chamber hyphema
- 4. Uncontrollable intraocular pressure
- 5. Zonular or capsular rupture
- 6. Bag-sulcus, sulcus-sulcus or unknown placement of the haptics
- 7. Suturing of incision required at time of surgery
- 8. Intraocular lens tilt or decentration
- 9. Significant sedation or retrobulbar block during surgery
- 10. Other procedure, such as pupil stretch, expanders, iris hooks during surgery

**Note:** Any subject in which surgery has been aborted for either eye should immediately be discontinued from the study and an exit form completed for that subject. These subjects will be followed up as per the clinic standard of care, monitored for safety, and their data will be excluded from the study efficacy analysis (obtained from FDA Database Research Results Feb, 05, 2009). All adverse events will be appropriately documented and reported.

Additionally, participants who are considered to be a vulnerable subject population are not to be enrolled into the study without prior written authorization from both the Sponsor and the IRB to ensure that a description of additional safeguards are in place during the consenting and enrollment processes. Vulnerable populations include, but are not limited to, the following:

- 1. Prisoners
- 2. Nursing home residents /institutionalized individuals
- 3. Mentally disabled /cognitively impaired individuals

6

- 4. Sponsor employees and their family members
- 5. Site employees and their family members that are directly and indirectly involved with the study
- 6. Students of the university or the principal investigator participating in the study
- 7. Economically and/or educationally disadvantaged individuals
- 8. Comatose individuals / traumatized individuals
- 9. Adults who do not read and/or write
- 10. Hearing impaired individuals
- 11. Terminally ill individuals / individuals with life-threatening conditions

#### 5. STUDY PROCEDURES

# 5.1. Informed Consent / Subject enrollment

Potential subjects will be identified from the patients presenting at the clinic. Additionally, a flyer will be placed in the check-in area of the different locations and on the practice website. Once identified as a study candidate, the patient will be asked if he/she would like to participate. The sub-investigator, study coordinator or an appropriately trained staff member will answer any and all questions and will obtain informed consent. A copy of the signed informed consent document will be given to the subject. The principal investigator will be available if the subject wants to discuss further details with him. Any testing that is part of the investigative site's standard preoperative cataract evaluation may be performed prior to the informed consent being signed, provided these tests are conducted within 90 days of surgery. The patient will understand that participation in the study, or declining to participate, will not affect his/her quality of care.

No subject will be enrolled into the study that does not meet the inclusion/exclusion criteria and does not sign the current approved informed consent document. Informed consent will be obtained prior to collecting any data for the study. The original signed documents will be maintained by the investigator as a permanent part of the subject's research records and a copy will be provided to the patient.

#### 5.2. Surgery Procedures:

Patients will receive either a non-toric or toric Vivity IOL based on the amount of astigmatism. The target refraction for the dominant eye will be plano ( $\pm 0.25$  D) and between -0.50 and -0.75 D (closest to -0.62) for the non-dominant eye.

# **5.3. Study Visit Schedule and Assessments** (Table 1).

#### **5.3.1.** Visit Schedule: Subjects will be examined at the following intervals:

- 1. Visit 1: Screening and enrollment: Preoperative evaluation completed not more than eight weeks before surgery
- 2. Visit 2: Day of Surgery for each eye
- 3. Visit 3: Month 3: 90 ±15 days postoperative after second eye surgery

#### 5.3.2. Measurements and evaluations

- 1. Visit 1: Informed consent process will be conducted at this visit. Assessments include best-corrected Snellen visual acuity, manifest refraction, intraocular pressure (IOP) using Goldman tonometer, slit lamp examination including dilated fundus exam, cataract density and type, and visual symptoms, patient satisfaction and spectacle independence questionnaires. Any testing that is part of the site's preoperative cataract surgery standard of care evaluation may be performed prior to signing the informed consent provided these tests are conducted within 90 days of the surgery and notation of the date performed is entered onto the CRF. The surgeon's standard pre-cataract surgery treatment will be used in all patients
- 2. Visit 2: The surgeon may use his preferred cataract extraction technique (manual or laser). The lens will be implanted in the bag. The following information will be captured the day of surgery: phaco technique (manual or laser), lens implanted and power, target refraction, residual astigmatism and axis for Barrett Toric Calculator (if applicable), additional surgical procedures, intraoperative complications, and any device deficiencies. The surgeon's standard post cataract surgery treatment will be used in all patients.

Visit 3: Slit lamp examination, manifest refraction, uncorrected as well as distance corrected visual acuities will be evaluated at 4 m, 66 cm and 40 cm and defocus curve, IOP, IOL orientation (if toric IOL and deem necessary by investigator), dilated fundus exam (as deem necessary by the investigator), visual symptoms, patient satisfaction and spectacle independence questionnaires, adverse events and any device deficiencies.

**Table 1**. Study Visit Schedule and Assessments

| | Visit 1<br>Screening | Visit 2 and 2A<br>DOS | Visit 3<br>3-Month<br>90 ±15 days |
|---|---|---|---|
| Informed Consent | X | | |
| Inclusion/Exclusion | X | X | |

CONFIDENTIAL CEP 20-002 Version 2.1 15Jun2020

| Demographics/PMH/Ocular | | | |
|-----------------------------------|---|---|-----|
| history | X | | |
| BCVA Snellen | Х | | |
| UCVA ETDRS (4m) | | | X* |
| UCIVA ETDRS (66 cm) | | | X** |
| UCNVA ETDRS (40 cm) | | | X** |
| Manifest refraction – Max Plus | | | Х |
| BCVA ETDRS (4m) target | | | Χ* |
| emmetropia | | | X** |
| DCIVA ETDRS (66 cm) target | | | Χ** |
| emmetropia | | | ^ |
| DCNVA ETDRS (40 cm) target | | | X** |
| emmetropia | | | ^ |
| Defocus curve target | | | X** |
| emmetropia | | | |
| BCVA ETDRS (4m) target | | | X* |
| nanovision | | | , , |
| DCIVA ETDRS (66 cm) target | | | X** |
| nanovision | | | |
| DCNVA ETDRS (40 cm) target | | | X** |
| nanovision Defects our to target | | | |
| Defocus curve target nanovision | | | X** |
| Intraocular Pressure (Goldman) | X | | X |
| SLE | X | | X |
| Dilated fundus exam | X | | χ† |
| | | | ^' |
| Cataract density / type | X | | |
| Toric IOL calculation | X | | |
| Intraoperative data | | Х | |
| Toric IOL position | | X | χ† |
| Questionnaires | X | | Х |
| AE/Device deficiencies | | X | Χ |

X To be performed as scheduled

<sup>\*</sup> Monocular and binocular testing

<sup>\*\*</sup> Binocular testing only

<sup>†</sup>To be performed as deem necessary by the investigator.

DC: distance corrected. DC, for the purpose of this study, is defined as corrected for the target refraction (i.e. emmetropia OU corrected for plano. Nanovison dominant eye corrected for plano and the non-dominant eye for -0.50).

9

#### 5.4. Study endpoint criteria

- 5.4.1. Patient Completion of Study: If a study patient has completed the final visit (Visit 3) of the study, he/she is considered to have completed the study.
- 5.4.2. Patient Discontinuation: Each study patient may voluntarily discontinue the study at any time they choose. Study patients who cannot complete the study for administrative reasons (e.g., non-compliance, failure to meet visit schedule, etc.) will be discontinued from the study. Study patients discontinued during the enrollment phase (prior to surgery) of the study will be replaced.
- 5.4.3. Patient Termination: A study patient will be terminated if the study patient develops any severe adverse event that may be related to the study. A study patient will receive appropriate treatment at the discretion of the investigator. Notification of termination will be clearly documented. These study patients are considered to have completed the study and will not be replaced.
- 5.4.4. Study Termination: The investigator with appropriate notification may terminate the study. If, after clinical observations, the investigator feels that it may be unwise to continue the study, he may stop the study.
- 5.4.5. Study Completion: The study will be complete when all enrolled patients have completed Visit 3 or have been terminated from the study.

#### 6. STATISTICAL CONSIDERATIONS

#### 6.1. Sample size

A total of 35 subjects will be enrolled. Browne suggests a general flat rule to 'use at least 30 subjects or greater to estimate a parameter'.

# 6.2. Statistical Analysis

All data will be collected by the site and entered into a database. Subjects will be assigned an ID number. Data analysis will be performed without patient identification. Statistical analysis will be performed using standard descriptive statistics and other tests as deemed appropriate based on the characteristics of the data to be analyzed. All

statistical tests will be two-sided and interpreted at a 5% significance level. Visual outcomes comparisons between the two targets (emmetropia and nanovision) will be made including cumulative visual acuity. Vision satisfaction, spectacle independence and visual symptoms will be compared to a historical control of patients implanted bilaterally with Vivity targeted for emmetropia OU. Data analysis will be conducted by a third-party consultant.

# 6.3. Safety Analyses

The type, severity, duration and frequency of reported ocular adverse events will be tabulated for each group. Adverse events will also be summarized for events that were considered treatment-related. Comparison of treatment groups with respect to the proportion of study patients reporting adverse events will be made using Fisher's Exact Test.

#### 7. DATA HANDLING AND RECORD KEEPING

# 7.1. Confidentiality

To ensure confidentiality in this study, records of the participants will be examined only by the principal investigator and research staff involved in the study. Study records will be kept on file. Any statistical analysis and publication will not include any subject identifiers. Medical records will be made available only for review by the investigators, Sponsor Company or Research Institution, the IRB, and other State or Federal Regulatory Agencies, if necessary. All information in these records will be kept confidential.

#### 7.2. Records Retention

The PI is accountable for the integrity, retention and security of all study related data. The investigator must maintain accurate, complete and current records relating to the clinical study. The investigator must maintain the required records during the investigation and for a period of 2 years after the date on which the investigation is terminated or completed then records will be scanned and kept electronically in a secured server.

#### 8. STUDY MONITORING, AUDITING, AND INSPECTING

The nature and location of all source documents will be identified to ensure that original data required to complete the case report forms (CRFs) exist and are accessible for verification. If electronic source records are maintained, these records must be 21 CFR Part 11 compliant and will be printed and certified for verification as needed.

Required examination must be recorded on the CRFs. CRFs will be used as source document. All data reported must have corresponding entries in the source documents. The principal investigator or sub-investigator must review the reported data and certify that the CRFs are

11

accurate and complete. No subject identifiers should be recorded on the CRFs beyond subject number, subject initials and study specific identifiers.

Data from CRFs will be entered into a database. Upon completion of the CRFs, the data will be reviewed by study designated personnel and statistician for accuracy and completeness. If corrections and/or any additions to the data are deemed necessary, queries will be generated. Designated research staff expected to respond to data queries in a timely manner and ensure that the corrections and changes made to the data in the database are reflected in the subjects' source documentation. Any changes will need to be initialed and dated by the authorized personnel making such changes.

Data will not be sold to third parties.

#### 9. INVESTIGATIONAL PRODUCT

#### 9.1. Description

Acrysof® IQ Vivity Intraocular Lens is a non-diffractive aspheric IOL that provides an extended range of vision maintaining low incidence of visual disturbances when compared to a monofocal IOL. The extended vision ranging from distance to near is obtained by a Wavefront-shaping technology on the anterior surface of the lens.

#### 9.2. Treatment/Dosing Regimen

The IOL will be implanted at time of uncomplicated routine cataract surgery. Intraocular lenses are implantable medical devices and are intended for long term use over the lifetime of the patient.

#### 9.3. Method for Assigning Subjects to Treatment/Dosing Groups

The statistician will provide randomization envelopes. The envelopes will be sequentially numbered.

# 9.4. Subject Compliance Monitoring

Since the IOL is implanted at time of cataract surgery, subject compliance will not be an issue in this particular study.

# 9.5. Packaging, Receiving, Storage, Dispensing and Return

N/A

#### **10. ETHICAL CONSIDERATIONS**

This clinical trial will be conducted in accordance with the principles of the Declaration of Helsinki, and Good clinical practice. The Investigator and all clinical trial staff will conduct the clinical trial in compliance with this protocol. The Investigator will ensure that all personnel

involved in the conduct of the clinical trial are qualified to perform their assigned duties through relevant education, training, and experience. Deviations from the clinical protocol must be documented in each subject's study records including the dates and reasons for each deviation. The PI must ensure that all aspects of the trial follow the applicable regulatory laws and conditions of approval imposed by the IRB.

#### 11. IN CASE OF AN INJURY RELATED TO THIS RESEARCH STUDY

Every effort to prevent study-related injury will be taken by the study doctor and staff. In the event a patient is injured as a direct result of the study while following the study instructions and requirements, the patient will be instructed to immediately contact the principal investigator and/or study staff. Treatment will be provided as needed for those injuries caused directly by this research study. In the event of injury or illness caused by or occurring during the participation in this study, all charges for medical care provided will be billed to the patient's insurance company. The medical care costs for injuries or illnesses that are not caused directly by the research study will not be covered.

# 12. CONFIDENTIALITY/PUBLICATION OF THE STUDY

The existence of this Study is confidential and should not be discussed with persons outside of the Study. Results will be submitted for publication and presentation at national and/or international meetings. A manuscript will be submitted to peer-review journals for publication but there is no guarantee of acceptance.